CLINICAL TRIAL: NCT00078338
Title: Phase IV, Multicenter, Open Label, Randomized Study of Rebif® 44 mcg Administered Three Times Per Week by Subcutaneous Injection Compared With Copaxone® 20 mg Administered Daily by Subcutaneous Injection in the Treatment of Relapsing Remitting Multiple Sclerosis
Brief Title: Rebif® Versus Copaxone® in the Treatment of Relapsing Remitting Multiple Sclerosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: EMD Serono (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24735
Record Dates: First submitted 2004-02-23; First posted 2004-02-26 (Estimated); Results first posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2017-09

CONDITIONS: Relapsing-remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1a; Glatiramer Acetate

ARMS (2):
- Rebif® (Experimental)
  Interventions: Drug: Rebif®
- Copaxone® (Active Comparator)
  Interventions: Drug: Copaxone®

INTERVENTIONS:
Drug: Rebif® — Subjects will be administered with Rebif® (Recombinant interferon beta-1a) as subcutaneous (SC) injection at a dose of 44 microgram (mcg) three times weekly (tiw).
  Other Names: Recombinant interferon beta-1a
  Arms: Rebif®
Drug: Copaxone® — Subjects will be administered with Copaxone® (Glatiramer acetate) as subcutaneous (SC) injection at a dose of 20 milligram (mg) once daily (qd).
  Other Names: Glatiramer acetate
  Arms: Copaxone®

SUMMARY:
The primary objective of the study is to assess the clinical efficacy of Rebif® 44 microgram (mcg) three times per week compared with Copaxone® 20 milligram (mg) daily in subjects with relapsing Multiple Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 60 years of age
* Have definite relapsing multiple sclerosis
* Have had one or more relapses within the prior 12 months
* Must be in a clinically stable or improving neurological state during the four weeks prior to Study Day 1
* Expanded Disability Status Scale (EDSS) score from 0 to 5.5, inclusive
* If female, she must either be post-menopausal or surgically sterilized; or use a hormonal contraceptive, intra uterine device, diaphragm with spermicide, or condom with spermicide, for the duration of the study; and be neither pregnant nor breast-feeding
* Confirmation that the subject is not pregnant must be established by a negative serum human chorionic gonadotropin (hCG) pregnancy test within 7 days of Study Day 1 and a negative urine pregnancy test on Study Day 1. A pregnancy test is not required if the subject is post-menopausal or surgically sterilized
* Be willing and able to comply with the protocol for the duration of the study
* Voluntarily provide written informed consent and, for USA sites only, a subject authorization under Health Insurance Portability and Accountability Act (HIPAA), prior to any study-related procedure that is not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to their future medical care

Exclusion Criteria:

* Have secondary progressive multiple sclerosis (SPMS) or primary progressive MS (PPMS)
* Prior use of any interferon or glatiramer acetate
* Have had treatment with oral or systemic corticosteroids or adrenocorticotrophic hormone (ACTH) within 4 weeks of Study Day 1 and within 7 days prior to the Day 1 magnetic resonance imaging (MRI)
* Have a psychiatric disorder that is unstable or would preclude safe participation in the study.
* Have significant leukopenia (white blood cell count < 0.5 times the lower limit of normal of the central laboratory) within 7 days of Study Day 1.
* Have elevated liver function tests (alanine aminotransferase [AST], aspartate aminotransferase [ALT], alkaline phosphatase > 2.0 times the upper limit of normal [ULN] of the central laboratory, or total bilirubin > 1.5 times the ULN of the central laboratory) within 7 days of Study Day 1 or a history of hepatitis (including infectious or drug-induced)
* Prior cytokine or anti-cytokine therapy within 3 months prior to Study Day 1
* Prior use of immunomodulatory or immunosuppressive therapy (including but not limited to cyclophosphamide, cyclosporin, methotrexate, azathioprine, linomide, mitoxantrone) within the 12 months prior to Study Day 1
* Prior use of cladribine or have received total lymphoid irradiation
* Have allergy or hypersensitivity to human serum albumin, mannitol, glatiramer acetate, natural or recombinant interferon-β, or any other components of the study drugs or gadolinium diethylenetriaminepentaacetic acid
* Have taken intravenous immunoglobulin or any other investigational drug or taken part in any experimental procedure in the 6 months prior to Study Day 1.
* Presence of systemic disease that might interfere with subject safety, compliance or evaluation of the condition under study (e.g. insulin-dependent diabetes, Lyme disease, clinically significant cardiac disease, human immunodeficiency virus [HIV], human T-cell lymphotrophic virus type I [HTLV-1])
* Have had plasma exchange in 3 months prior to Study Day 1.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 764 (Actual)
Dates: Start 2004-02-16 (Actual); Primary Completion 2006-11-28 (Actual); Study Completion 2006-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (80):
- United States (41):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Barrow Neurology Clinics, Phoenix, Arizona
  - Northwest NeuroSpecialists, Tucson, Arizona
  - University of California, Davis, Sacramento, California
  - Kaiser Permanente Neurology, San Diego, California
  - Advanced Neurology of Colorado, LLC, Fort Collins, Colorado
  - The MS Treatment Center at Griffin Hospital, Derby, Connecticut
  - Associated Neurologists of Southern Connecticut, P.C., Fairfield, Connecticut
  - Neurological Center of South Florida, Miami, Florida
  - Harbourside Medical Plaza, Tampa, Florida
  - Shepherd Center, Atlanta, Georgia
  - University Chicago Hospitals, Chicago, Illinois
  - Consultants In Neurology, Ltd., Northbrook, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - University of Maryland MD Center for MS, Baltimore, Maryland
  - University Of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Henry Ford Hospital Dept of Neurology, Detroit, Michigan
  - The Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - University of Minnesota Medical School, Dept of Neurology, Minneapolis, Minnesota
  - Nevada Neurological Consultants, Henderson, Nevada
  - Albany Medical College Dept of Neurology MC-70, Albany, New York
  - Neurology University of Rochester, Rochester, New York
  - SUNY At Stony Brook U Hospital - Department of Neurology, Stony Brook, New York
  - SUNY Upstate Medical University Dept of Neurology, Syracuse, New York
  - MS Center/CHS, Charlotte, North Carolina
  - Wake Forest Univ. Health Sciences, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - Oak Clinic for Multiple Sclerosis, Uniontown, Ohio
  - Medford Neurological and Spine Clinic, Medford, Oregon
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Physicians Dept of Neurology, Philadelphia, Pennsylvania
  - Baptist West Hospital, Knoxville, Tennessee
  - University of Texas-Houston, Houston, Texas
  - Central Texas Neurology, Round Rock, Texas
  - Neurology Health Care Service / Fletcher Allen Health Care, Burlington, Vermont
  - Neurology Center of Fairfax, Fairfax, Virginia
  - Blue Ridge Research Center, Roanoke, Virginia
  - Minor & James Medical, PLLC, Seattle, Washington
  - CAMC Institute, Charleston, West Virginia
  - Center for Neurological Disorders, Milwaukee, Wisconsin
- Argentina (6):
  - Servicio de Neurologia, Buenos Aires
  - Departmento Enfermedades Desmielinizantes, Buenos Aires
  - Servicio de Neurologia Departmento Enfermedades Desmielinizantes, Buenos Aires
  - Seccion Neurolgia Instituto INEBA, Buenos Aires
  - Fundacion Rosarina de Neurorehabilitacion, Rosario
  - Dept Neurologia Sanatorio Britanico de Rosario, Rosario
- OO Landes-Nervenklinik, Linz, Austria
- Campus Ribeirao Preto Faculdade de Medicina de Sao Paolo, Riberao Preto-SP, Brazil
- France (2):
  - Dept of Neurology CHU Timone, Marseille
  - Hopital Pontchaillou, Rennes
- Germany (2):
  - Dept of Neurology Johannes Gutenberg University, Mainz
  - Dept of Neurology Universitatsklinikum Munster, Münster
- Italy (4):
  - Dept of Neurological and Psychiatric Sciences University of Bari, Bari
  - Dept of Neurosciences Oftamology and Genetics Univ of Genoa, Genoa
  - Dept Neurology Ospedale San Raffaele, Milan
  - Dept of Neurological Sciences University La Sapienza Rome, Rome
- Netherlands (2):
  - Academisch Ziekenhuis Vrije Universiteit, Amsterdam
  - MS Center Nijmegen, Nijmegen
- Russia (11):
  - City Clinical Hospital No 83, Moscow
  - Dept Of Neurology and Neurosurgery, Russian State Med Univ, Moscow
  - State Instituion Central Clinical Milatary Hospital, Moscow
  - Scientific Research Center of Neurology Russian MOH, Moscow
  - Department of Neurology City Hospital #33, Nizhny Novgorod
  - Institute of Clinical Immunology RAMS, Novosibirsk
  - Military Medical Academy, Saint Petersburg
  - Dept of Neurology St Petersburg State Medical University, Saint Petersburg
  - Dept of MS Institute for Human Brain of R.A.Sci, Saint Petersburg
  - Dept of Neurology Medical Clinic of Russian MoH, Saint Petersburg
  - Chair of Nuerological Diseases and Medical Genetics, Yaroslavl
- Spain (4):
  - Neuroinmunologia Clinica Hospital Vall d'Hebron, Barcelona
  - Servicio de Neurologia Hospital Bellvitge, L'Hospitalet de Llobregat
  - Neurologia Hospital Carlos Haya, Málaga
  - Unidad de EM Neurologia Hospital Virgen Macarena, Seville
- Dept Of Neurology, Zurich, Switzerland
- United Kingdom (5):
  - Department of Neurology, Whitechapel, London
  - Department Of Neurology Royal London Hospital, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Div of Clinical Neurology B Floor Medical School Univ Hospital, Nottingham
  - Division of Clinical Neurology Medical School Universtity Hopsital, Nottingham

REFERENCES:
- [Result] Mikol DD, Barkhof F, Chang P, Coyle PK, Jeffery DR, Schwid SR, Stubinski B, Uitdehaag B; REGARD study group. Comparison of subcutaneous interferon beta-1a with glatiramer acetate in patients with relapsing multiple sclerosis (the REbif vs Glatiramer Acetate in Relapsing MS Disease [REGARD] study): a multicentre, randomised, parallel, open-label trial. Lancet Neurol. 2008 Oct;7(10):903-14. doi: 10.1016/S1474-4422(08)70200-X. Epub 2008 Sep 11. PMID 18789766

RESULTS

PARTICIPANT FLOW:
Groups:
- Rebif®: Subjects were administered with Rebif® (Recombinant interferon beta-1a) as subcutaneous (SC) injection at a dose of 44 microgram (mcg) three times weekly (tiw).
- Copaxone®: Subjects were administered with Copaxone® (Glatiramer acetate) as subcutaneous (SC) injection at a dose of 20 milligram (mg) once daily (qd).
Period: Overall Study
Arm/Group | Rebif® | Copaxone®
Started | 386 | 378
Safety Population | 381 (Safety population=subjects who received at least 1 dose of treatment and had followup safety data.) | 375 (Safety population=subjects who received at least 1 dose of treatment and had followup safety data.)
Completed | 301 | 324
Not Completed | 85 | 54
Not completed — Adverse Event | 31 | 24
Not completed — Lost to Follow-up | 17 | 2
Not completed — Protocol Violation | 2 | 2
Not completed — Disease Progression | 4 | 7
Not completed — Other | 28 | 16
Not completed — Subjects randomized, but not treated | 3 | 3

BASELINE CHARACTERISTICS:
Population: The intent to treat (ITT) population consisted of all subjects who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rebif® | Copaxone® | Total
Number analyzed (Participants) | 386 | 378 | 764
Age, Customized [Number; unit: Participants]
  Less than 18 years | 0 | 0 | 0
  18 years to 64 years | 386 | 378 | 764
  Greater than 64 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 267 | 272 | 539
  Male | 119 | 106 | 225

OUTCOME MEASURES:

1. Primary Outcome: Time to First Relapse
Description: Relapse was defined as new, worsening or recurrent neurological symptoms attributed to multiple sclerosis that last for at least 24 hours without fever or infection, or adverse reaction to prescribed medication, preceded by a stable or improving neurological status of at least 30 days. These new or worsening symptoms should be noted by subject and must be accompanied by at least 1 of the following: An increase of greater than or equal to (>=) 1 grade in >=2 functional scales of the Expanded Disability Status Scale (EDSS) or an increase of >=2 grades in 1 functional scale of the EDSS or an increase of >= 0.5 or an increase of >=1.0 in EDSS if the previous EDSS was 0. Time to first relapse was defined as the time in days from the date of first dose of study treatment to the date of first multiple sclerosis relapse. The mean time to first relapse for the 25th percentile and the 30th percentile during the 96-week treatment period was measured by Kaplan-Meier estimates and was reported.
Time Frame: Baseline up to 96 weeks
Population: The ITT population consisted of all subjects who were randomized.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rebif® | Copaxone®
Number analyzed (Participants) | 386 | 378
days
  25th Percentile | 332.0 (10.9) | 290.0 (9.5)
  30th Percentile | 495.0 (16.3) | 432.0 (14.2)
Statistical Analysis 1: Comparison: Rebif® vs Copaxone®; Test type: Superiority or Other; p = 0.643, Cox proportional hazards model; Hazard Ratio (HR) = 0.943, 95% CI 2-sided [0.74 to 1.21]

ADVERSE EVENTS:
Description: The Safety population consisted of all subjects who received at least 1 dose of study treatment and had follow-up safety data.
Arm/Group | Rebif® | Copaxone®
Serious Adverse Events (participants affected / at risk) | 29/381 | 27/375
Other Adverse Events (participants affected / at risk) | 346/381 | 320/375
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rebif® (N=381) | Copaxone® (N=375)
Acute sinusitis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1
Dental caries (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Postoperative infection (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 2
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Jejunal perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Salivary gland cyst (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 2 | 1
Face oedema (General disorders) | 0 | 2
Adverse drug reaction (General disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Depression (Psychiatric disorders) | 2 | 1
Affective disorder (Psychiatric disorders) | 1 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 0
Delusional disorder, persecutory type (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1
Paranoia (Psychiatric disorders) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Haemochromatosis (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rebif® (N=381) | Copaxone® (N=375)
Injection site erythema (General disorders) | 121 | 114
Influenza like illness (General disorders) | 119 | 5
Headache (Nervous system disorders) | 74 | 35
Injection site pain (General disorders) | 47 | 53
Injection site pruritus (General disorders) | 8 | 75
Nasopharyngitis (Infections and infestations) | 34 | 44
Injection site bruising (General disorders) | 33 | 38
Nausea (Gastrointestinal disorders) | 25 | 28
Depression (Psychiatric disorders) | 30 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 25 | 26
Sinusitis (Infections and infestations) | 18 | 29
Injection site swelling (General disorders) | 4 | 42
Upper respiratory tract infection (Infections and infestations) | 15 | 27
Influenza (Infections and infestations) | 18 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 22
Urinary tract infection (Infections and infestations) | 17 | 20
Pyrexia (General disorders) | 23 | 14
Injection site induration (General disorders) | 9 | 25
Anxiety (Psychiatric disorders) | 21 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 22 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 22
Alanine aminotransferase increased (Investigations) | 21 | 5
Adverse drug reaction (General disorders) | 0 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other